CLINICAL TRIAL: NCT06822322
Title: The European Bifurcation Club Randomized Trial of Stepwise Provisional Stenting Versus Drug Coated Balloon Therapy for Non-left Main True Coronary Bifurcations - EBC DCB Study
Brief Title: The European Bifurcation Club Randomized Trial of Stepwise Provisional Stenting Versus Drug Coated Balloon Therapy for Non-left Main True Coronary Bifurcations
Acronym: EBC DCB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ceric Sàrl (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EBC DCB
Record Dates: First submitted 2025-01-23; First posted 2025-02-12 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease (non-left Main); Coronary Bifurcation Lesion
Keywords: non-left coronary bifurcation; drug coated balloon; drug eluted stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Angioplasty, Balloon, Coronary

STUDY DESIGN:
Intervention Model Description: Post-market study to compare Drug Coated Balloon versus Drug Eluted Stent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stepwise Provisional Stent Strategy (Active Comparator): Coronary guide wires are passed into both the main vessel (MV) and side branch (SB). Stenting of the MV is undertaken with a wire jailed in the SB to preserve SB flow and access. Stent diameter is chosen according to the diameter of the distal MV. Following stent deployment, the stent portion in the proximal MV is dilated with a short non-compliant balloon (POT technique) to achieve full expansion and apposition.
  Finally, after POT technique, SB is rewired and a kissing balloon inflation (KBI) is undertaken to address any plaque or carina shift and to open stent struts. Thus, non-compliant balloons sized to the diameter of the distal MV and SB are sequentially inflated at high pressure, and then simultaneously at low pressure.
  Further SB treatment is required only if <TIMI 3 flow, significant stenosis >70% or significant dissection. Thus, a side vessel stent implantation followed with KBI are mandatory.
  Interventions: Procedure: Percutaneous Coronary Angioplasty; Device: Stepwise Provisional Stent Strategy
- Drug Coated Balloon Strategy (Experimental): Coronary guide wires are passed into both the main vessel (MV) and side branch (SB). If residual stenosis remains >30%, or TIMI flow<3, or dissection propagation, the stenting of the MV is mandatory.
  Otherwise, a paclitaxel-drug coated balloon (DCB) is inflated in the prepared SB for 60 seconds at nominal pressure.
  If residual stenosis remains >50%, or TIMI flow<3, or dissection propagation, the operator will decide between prolonged balloon dilatation (1-2 minutes) or stent implantation, in the SB.
  After SB treatment, MV is treated with a DCB at nominal pressure only, sized 1:1 with the proximal MV, for 60 seconds. If result is unacceptable, MV stenting followed with kissing balloon inflation and DCB or stent implantation into SB, are mandatory.
  The procedure is complete when the MV has residual stenosis <30%, has TIMI 3 flow and has no dissection propagation ; when the SB has residual stenosis <50%, has TIMI 3 flow and has no dissection propagation.
  Interventions: Procedure: Percutaneous Coronary Angioplasty; Device: Drug Coated Balloon Strategy; Device: Cross-Over Stepwise Provisional Stent Strategy

INTERVENTIONS:
Procedure: Percutaneous Coronary Angioplasty — A Percutaneous Coronary Intervention is used in both arms, with the drug Zotarolimus for stenting strategy and Paclitaxel for balloon strategy.
  Coronary guide wires are passed into both the distal main vessel (distal MV) and side branch (SB) and predilation of MV on a 1:1 basis is required.
  The device component dilates the vessel lumen by Percutaneous Transluminal Coronary Angioplasty (PTCA), while the drug is intended to reduce the proliferative response associated with restenosis.
Device: Stepwise Provisional Stent Strategy — In the stepwise provisional stent strategy, stenting of the MV is undertaken with a wire jailed in the SB. Then, non-compliant balloons sized to the diameter of the distal MV and SB are sequentially inflated at high pressure, and then simultaneously at low pressure (kissing balloon inflation ; KBI).
  Arms: Stepwise Provisional Stent Strategy
Device: Drug Coated Balloon Strategy — In the drug coated balloon (DCB) strategy, SB is prepared with a balloon at a 1:1 diameter, followed with a 1:1 sized DCB inflation for 60 seconds at nominal pressure. Then, MV is re-evaluated and treated with DCB at nominal pressure only, sized 1:1 with the proximal MV, for 60 seconds.
  Arms: Drug Coated Balloon Strategy
Device: Cross-Over Stepwise Provisional Stent Strategy — Following Drug Coated Balloon treatment in the Main vessel (MV) in the Drug Coated Balloon Arm, if the result is unacceptable in the MV, with either TIMI>3 flow and/or dissection propagation, MV stenting is mandatory followed with Kissing Balloon Inflation (KBI), where non-compliant balloons sized to the diameter of the distal main and side branch are sequentially inflated at high pressure, and then simultaneously at low pressure. If the cross-over stent implantation in the MV is used, a further SB treatment with either DCB or stent implantation is used, according to operator preference.
  Arms: Drug Coated Balloon Strategy

SUMMARY:
Clinical outcomes are worse in patients with coronary artery bifurcation lesions, even if commonly encountered in clinical practice. The use of drug coated balloons within bifurcation lesions offers the acute advantage of a more straightforward procedure, without recrossing and deformation of a stent. Thus, the primary objective of this study is to determine if Drug Coated Balloon treatment of non-left main true coronary artery bifurcation lesions is non-inferior (similar) to a provisional strategy with Drug Eluted Stent deployment.

DETAILED DESCRIPTION:
The EBC DCB study is an investigator-initiated, prospective, multi-centre, open-label, randomized (1:1) non-inferiority trial.

Patients with non-left main bifurcations requiring revascularisation and both the main vessel and side branch significantly diseased ( ≥2.5mm and Medina 1/1/1, 1/0/1 or 0/1/1), constitute the source population. Patients with no more than two additional coronary disease may be considered for the study, with only one bifurcation lesion included.

Patients, pre-selected by their referring physicians, will be screened for eligibility by the study team. If patients fulfill all inclusion and do not meet exclusion criteria, they will be informed about the study's purpose and course and will be asked for participation and written informed consent. 20 sites will be involved, in 7 European countries and South Korea, for a total of 750 patients. After a 2-years recruitment period, the trial will include a Follow-Up period at 6-months, 1-year, 3-years, 5-years and 8-years. The 1-year check point will constitute the primary endpoint where the Bifurcation Orientated Composite Endpoint (BOCE) will be analyzed for non-inferiority (further analysis for superiority, if non-inferiority met).

ELIGIBILITY:
Inclusion Criteria:

* True non-left main bifurcation disease with both MV and SB involvement (i.e Medina 1/1/1, 1/0/1, 0/1/1)
* Bifurcation lesion responsible for an acute or chronic coronary syndrome with at least one of the following:

  * ≥70% angiographic MV and SB diameter stenosis
  * Positive non-invasive testing for ischaemia
  * Positive coronary physiology for ischaemia
* Significant SB as described by diameter stenosis ≥50% and all of the following:

  * SB length ≥73mm
  * SB diameter ≥2.5mm
  * Absence of another SB emerging distally from the MV
  * Non-dominant circumflex artery, if SB is a diagonal branch.

Exclusion criteria

* Patients <18 years old
* STEMI <48 hours
* Cardiogenic shock
* Chronic total occlusion involving target bifurcation vessels
* In-stent restenosis
* Patient life expectancy <12 months
* >2 other coronary lesions (target or non-target) planned for treatment
* SYNTAX score >32
* Platelet count ≤50x109/mm3
* Left ventricular ejection fraction ≤20%
* Participation in another investigational drug or device study
* Patient unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2035-08 (Estimated)

PRIMARY OUTCOMES:
Bifurcation Orientated Composite Endpoint (BOCE) | At 1-year, after the day of enrollment
  The BOCE is defined by:
  * cardiovascular death,
  * target bifurcation-related myocardial infarction or
  * target bifurcation revascularisation

SECONDARY OUTCOMES:
Bifurcation Orientated Composite Endpoint (BOCE) | At 3, 5 and 8-years
  BOCE non-inferiority and superiority
Individual components of the Primary Endpoint | At 1, 3, 5 and 8-years
  * cardiovascular death
  * target bifurcation-related myocardial infarction
  * target bifurcation revascularisation
Safety Composite Endpoint | At 1, 3, 5 and 8-years
  - Safety Composite Endpoint defined as:
  * BARC bleeding (2/3/5)
  * Definite stent/lesion thrombosis
  * Stroke
  * MI
  * All-cause mortality
Individual components of the Safety Composite Endpoint | At 1, 3, 5 and 8-years
  * BARC bleeding (2/3/5)
  * Definite stent/lesion thrombosis
  * Stroke
  * MI
  * All-cause mortality
BARC 3 or 5 bleeding rate | At 1, 3, 5 and 8-years
  BARC 3 or 5 bleeding rate
Angina status | At 1, 3, 5 and 8-years
  Questionnaire: Seattle Angina Questionnaire - 7 (SAQ-7) Scale Range (Minimum and Maximum Values): 0 to 100 Higher scores indicate a better outcome (better health status, less angina, and better quality of life).
Angina index | At 1, 3, 5 and 8-years
  No. of antianginals

CONTACTS AND LOCATIONS:
Overall Officials: David HILDICK-SMITH, Prof., MD, Principal Investigator — Brighton & Sussex University NHS Hospitals Trust - Royal Sussex County Hospital - Eastern Road - Brighton, East Sussex - BN25BE, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jeger RV, Farah A, Ohlow MA, Mangner N, Mobius-Winkler S, Leibundgut G, Weilenmann D, Wohrle J, Richter S, Schreiber M, Mahfoud F, Linke A, Stephan FP, Mueller C, Rickenbacher P, Coslovsky M, Gilgen N, Osswald S, Kaiser C, Scheller B; BASKET-SMALL 2 Investigators. Drug-coated balloons for small coronary artery disease (BASKET-SMALL 2): an open-label randomised non-inferiority trial. Lancet. 2018 Sep 8;392(10150):849-856. doi: 10.1016/S0140-6736(18)31719-7. Epub 2018 Aug 28. PMID 30170854
- [Background] Ellis SG, Kereiakes DJ, Metzger DC, Caputo RP, Rizik DG, Teirstein PS, Litt MR, Kini A, Kabour A, Marx SO, Popma JJ, McGreevy R, Zhang Z, Simonton C, Stone GW; ABSORB III Investigators. Everolimus-Eluting Bioresorbable Scaffolds for Coronary Artery Disease. N Engl J Med. 2015 Nov 12;373(20):1905-15. doi: 10.1056/NEJMoa1509038. Epub 2015 Oct 12. PMID 26457558
- [Background] Hildick-Smith D, Behan MW, Lassen JF, Chieffo A, Lefevre T, Stankovic G, Burzotta F, Pan M, Ferenc M, Bennett L, Hovasse T, Spence MJ, Oldroyd K, Brunel P, Carrie D, Baumbach A, Maeng M, Skipper N, Louvard Y. The EBC TWO Study (European Bifurcation Coronary TWO): A Randomized Comparison of Provisional T-Stenting Versus a Systematic 2 Stent Culotte Strategy in Large Caliber True Bifurcations. Circ Cardiovasc Interv. 2016 Sep;9(9):e003643. doi: 10.1161/CIRCINTERVENTIONS.115.003643. PMID 27578839
- [Background] Hildick-Smith D, de Belder AJ, Cooter N, Curzen NP, Clayton TC, Oldroyd KG, Bennett L, Holmberg S, Cotton JM, Glennon PE, Thomas MR, Maccarthy PA, Baumbach A, Mulvihill NT, Henderson RA, Redwood SR, Starkey IR, Stables RH. Randomized trial of simple versus complex drug-eluting stenting for bifurcation lesions: the British Bifurcation Coronary Study: old, new, and evolving strategies. Circulation. 2010 Mar 16;121(10):1235-43. doi: 10.1161/CIRCULATIONAHA.109.888297. Epub 2010 Mar 1. PMID 20194880
- [Background] Konishi H, Habara M, Nasu K, Koshida R, Kinoshita Y, Tsuchikane E, Terashima M, Matsubara T, Suzuki T. Impact of Optimal Preparation Before Drug-Coated Balloon Dilatation for De Novo Lesion in Patients With Coronary Artery Disease. Cardiovasc Revasc Med. 2022 Feb;35:91-95. doi: 10.1016/j.carrev.2021.03.012. Epub 2021 Mar 20. PMID 33766488
- [Background] Jeger RV, Eccleshall S, Wan Ahmad WA, Ge J, Poerner TC, Shin ES, Alfonso F, Latib A, Ong PJ, Rissanen TT, Saucedo J, Scheller B, Kleber FX; International DCB Consensus Group. Drug-Coated Balloons for Coronary Artery Disease: Third Report of the International DCB Consensus Group. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1391-1402. doi: 10.1016/j.jcin.2020.02.043. Epub 2020 May 27. PMID 32473887
- [Background] Ninomiya K, Serruys PW, Colombo A, Reimers B, Basavarajaiah S, Sharif F, Testa L, Di Mario C, Nerla R, Ding D, Huang J, Kotoku N, Kageyama S, Kageyama M, Sevestre E, Fezzi S, Dijkstra J, O'Leary N, Morel MA, Garg S, Cortese B, Onuma Y. A Prospective Randomized Trial Comparing Sirolimus-Coated Balloon With Paclitaxel-Coated Balloon in De Novo Small Vessels. JACC Cardiovasc Interv. 2023 Dec 11;16(23):2884-2896. doi: 10.1016/j.jcin.2023.09.026. Epub 2023 Oct 23. PMID 37877914
- [Background] Latib A, Agostoni P, Dens J, Patterson M, Lancellotti P, Tam FCC, Schotborgh C, Kedhi E, Stella P, Shen C, Wetzels G, Testa L; PREVAIL Study Investigators. Paclitaxel Drug-Coated Balloon for the Treatment of De Novo Small-Vessel and Restenotic Coronary Artery Lesions: 12-Month Results of the Prospective, Multicenter, Single-Arm PREVAIL Study. J Invasive Cardiol. 2021 Nov;33(11):E863-E869. doi: 10.25270/jic/21.00119. Epub 2021 Aug 19. PMID 34433695
- [Background] Widder JD, Cortese B, Levesque S, Berliner D, Eccleshall S, Graf K, Doutrelant L, Ahmed J, Bressollette E, Zavalloni D, Piraino D, Roguin A, Scheller B, Stella PR, Bauersachs J. Coronary artery treatment with a urea-based paclitaxel-coated balloon: the European-wide FALCON all-comers DCB Registry (FALCON Registry). EuroIntervention. 2019 Jul 20;15(4):e382-e388. doi: 10.4244/EIJ-D-18-00261. PMID 29992902
- [Background] Latib A, Colombo A, Castriota F, Micari A, Cremonesi A, De Felice F, Marchese A, Tespili M, Presbitero P, Sgueglia GA, Buffoli F, Tamburino C, Varbella F, Menozzi A. A randomized multicenter study comparing a paclitaxel drug-eluting balloon with a paclitaxel-eluting stent in small coronary vessels: the BELLO (Balloon Elution and Late Loss Optimization) study. J Am Coll Cardiol. 2012 Dec 18;60(24):2473-80. doi: 10.1016/j.jacc.2012.09.020. Epub 2012 Nov 14. PMID 23158530
- [Background] Gao XF, Ge Z, Kan J, Kong XQ, Wang Y, Qiu CG, Tresukosol D, He YQ, Wu Q, Li JF, Yuan HT, Shen C, Chen X, Munawar M, Hanif B, Santoso T, Shin ES, Sheiban I, Ye F, Zhang JJ, Chen SL; DCB-BIF investigators. Rationale and design for comparison of non-compliant balloon with drug-coating balloon angioplasty for side branch after provisional stenting for patients with true coronary bifurcation lesions: a prospective, multicentre and randomised DCB-BIF trial. BMJ Open. 2022 Mar 11;12(3):e052788. doi: 10.1136/bmjopen-2021-052788. PMID 35277400
- [Background] Kleber FX, Rittger H, Ludwig J, Schulz A, Mathey DG, Boxberger M, Degenhardt R, Scheller B, Strasser RH. Drug eluting balloons as stand alone procedure for coronary bifurcational lesions: results of the randomized multicenter PEPCAD-BIF trial. Clin Res Cardiol. 2016 Jul;105(7):613-21. doi: 10.1007/s00392-015-0957-6. Epub 2016 Jan 14. PMID 26768146
- [Background] Bruch L, Zadura M, Waliszewski M, Platonic Z, Eranen J, Scheller B, Gotting B, Herberger D, Palmieri C, Sinicropi G, Motz W. Results From the International Drug Coated Balloon Registry for the Treatment of Bifurcations. Can a Bifurcation Be Treated Without Stents? J Interv Cardiol. 2016 Aug;29(4):348-56. doi: 10.1111/joic.12301. Epub 2016 May 31. PMID 27242273
- [Background] Schulz A, Hauschild T, Kleber FX. Treatment of coronary de novo bifurcation lesions with DCB only strategy. Clin Res Cardiol. 2014 Jun;103(6):451-6. doi: 10.1007/s00392-014-0671-9. Epub 2014 Feb 14. PMID 24522798
- [Background] Vos NS, Fagel ND, Amoroso G, Herrman JR, Patterson MS, Piers LH, van der Schaaf RJ, Slagboom T, Vink MA. Paclitaxel-Coated Balloon Angioplasty Versus Drug-Eluting Stent in Acute Myocardial Infarction: The REVELATION Randomized Trial. JACC Cardiovasc Interv. 2019 Sep 9;12(17):1691-1699. doi: 10.1016/j.jcin.2019.04.016. Epub 2019 May 21. PMID 31126887
- [Background] Jeger RV, Farah A, Ohlow MA, Mangner N, Mobius-Winkler S, Weilenmann D, Wohrle J, Stachel G, Markovic S, Leibundgut G, Rickenbacher P, Osswald S, Cattaneo M, Gilgen N, Kaiser C, Scheller B; BASKET-SMALL 2 Investigators. Long-term efficacy and safety of drug-coated balloons versus drug-eluting stents for small coronary artery disease (BASKET-SMALL 2): 3-year follow-up of a randomised, non-inferiority trial. Lancet. 2020 Nov 7;396(10261):1504-1510. doi: 10.1016/S0140-6736(20)32173-5. Epub 2020 Oct 19. PMID 33091360
- [Background] Cortese B, Testa G, Rivero F, Erriquez A, Alfonso F. Long-Term Outcome of Drug-Coated Balloon vs Drug-Eluting Stent for Small Coronary Vessels: PICCOLETO-II 3-Year Follow-Up. JACC Cardiovasc Interv. 2023 May 8;16(9):1054-1061. doi: 10.1016/j.jcin.2023.02.011. Epub 2023 Apr 19. PMID 37164603
- [Background] Megaly M, Buda K, Saad M, Tawadros M, Elbadawi A, Basir M, Abbott JD, Rinfret S, Alaswad K, Brilakis ES. Outcomes With Drug-Coated Balloons vs. Drug-Eluting Stents in Small-Vessel Coronary Artery Disease. Cardiovasc Revasc Med. 2022 Feb;35:76-82. doi: 10.1016/j.carrev.2021.03.008. Epub 2021 Mar 20. PMID 33858783
- [Background] Jing QM, Zhao X, Han YL, Gao LL, Zheng Y, Li ZQ, Yang P, Cong HL, Gao CY, Jiang TM, Li H, Li JX, Wang DM, Wang G, Cong ZC, Zhang Z. A drug-eluting Balloon for the trEatment of coronarY bifurcatiON lesions in the side branch: a prospective multicenter ranDomized (BEYOND) clinical trial in China. Chin Med J (Engl). 2020 Apr 20;133(8):899-908. doi: 10.1097/CM9.0000000000000743. PMID 32265425
- [Background] Herrador JA, Fernandez JC, Guzman M, Aragon V. Drug-eluting vs. conventional balloon for side branch dilation in coronary bifurcations treated by provisional T stenting. J Interv Cardiol. 2013 Oct;26(5):454-62. doi: 10.1111/joic.12061. PMID 24106744
- [Background] Lopez Minguez JR, Nogales Asensio JM, Doncel Vecino LJ, Sandoval J, Romany S, Martinez Romero P, Fernandez Diaz JA, Fernandez Portales J, Gonzalez Fernandez R, Martinez Caceres G, Merchan Herrera A, Alfonso Manterola F; BABILON Investigators. A prospective randomised study of the paclitaxel-coated balloon catheter in bifurcated coronary lesions (BABILON trial): 24-month clinical and angiographic results. EuroIntervention. 2014 May;10(1):50-7. doi: 10.4244/EIJV10I1A10. PMID 24832638
- [Background] Radke PW, Joner M, Joost A, Byrne RA, Hartwig S, Bayer G, Steigerwald K, Wittchow E. Vascular effects of paclitaxel following drug-eluting balloon angioplasty in a porcine coronary model: the importance of excipients. EuroIntervention. 2011 Oct 30;7(6):730-7. doi: 10.4244/EIJV7I6A116. PMID 21986331
- [Background] Posa A, Nyolczas N, Hemetsberger R, Pavo N, Petnehazy O, Petrasi Z, Sangiorgi G, Gyongyosi M. Optimization of drug-eluting balloon use for safety and efficacy: evaluation of the 2nd generation paclitaxel-eluting DIOR-balloon in porcine coronary arteries. Catheter Cardiovasc Interv. 2010 Sep 1;76(3):395-403. doi: 10.1002/ccd.22468. PMID 20839356
- [Background] Belkacemi A, Agostoni P, Voskuil M, Stella PR. Coronary bifurcation lesions treated with the drug-eluting balloon: a preliminary insight from the DEBIUT study. EuroIntervention. 2011 May;7 Suppl K:K66-9. doi: 10.4244/EIJV7SKA12. PMID 22027731
- [Background] Stella PR, Belkacemi A, Dubois C, Nathoe H, Dens J, Naber C, Adriaenssens T, van Belle E, Doevendans P, Agostoni P. A multicenter randomized comparison of drug-eluting balloon plus bare-metal stent versus bare-metal stent versus drug-eluting stent in bifurcation lesions treated with a single-stenting technique: six-month angiographic and 12-month clinical results of the drug-eluting balloon in bifurcations trial. Catheter Cardiovasc Interv. 2012 Dec 1;80(7):1138-46. doi: 10.1002/ccd.23499. Epub 2012 Mar 15. PMID 22422607
- [Background] Berland J, Lefevre T, Brenot P, Fajadet J, Motreff P, Guerin P, Dupouy P, Schandrin C; DEBSIDE trial investigators. DANUBIO - a new drug-eluting balloon for the treatment of side branches in bifurcation lesions: six-month angiographic follow-up results of the DEBSIDE trial. EuroIntervention. 2015 Dec;11(8):868-76. doi: 10.4244/EIJV11I8A177. PMID 26696455
- [Background] Jim MH, Lee MK, Fung RC, Chan AK, Chan KT, Yiu KH. Six month angiographic result of supplementary paclitaxel-eluting balloon deployment to treat side branch ostium narrowing (SARPEDON). Int J Cardiol. 2015;187:594-7. doi: 10.1016/j.ijcard.2015.04.002. Epub 2015 Apr 2. No abstract available. PMID 25863309
- [Background] Worthley S, Hendriks R, Worthley M, Whelan A, Walters DL, Whitbourn R, Meredith I. Paclitaxel-eluting balloon and everolimus-eluting stent for provisional stenting of coronary bifurcations: 12-month results of the multicenter BIOLUX-I study. Cardiovasc Revasc Med. 2015 Oct-Nov;16(7):413-7. doi: 10.1016/j.carrev.2015.07.009. Epub 2015 Aug 10. PMID 26346023
- [Background] Mathey DG, Wendig I, Boxberger M, Bonaventura K, Kleber FX. Treatment of bifurcation lesions with a drug-eluting balloon: the PEPCAD V (Paclitaxel Eluting PTCA Balloon in Coronary Artery Disease) trial. EuroIntervention. 2011 May;7 Suppl K:K61-5. doi: 10.4244/EIJV7SKA11. PMID 22027730
- [Background] Bocci G, Di Paolo A, Danesi R. The pharmacological bases of the antiangiogenic activity of paclitaxel. Angiogenesis. 2013 Jul;16(3):481-92. doi: 10.1007/s10456-013-9334-0. Epub 2013 Feb 7. PMID 23389639
- [Background] Her AY, Ann SH, Singh GB, Kim YH, Okamura T, Garg S, Koo BK, Shin ES. Serial Morphological Changes of Side-Branch Ostium after Paclitaxel-Coated Balloon Treatment of De Novo Coronary Lesions of Main Vessels. Yonsei Med J. 2016 May;57(3):606-13. doi: 10.3349/ymj.2016.57.3.606. PMID 26996558
- [Background] Kitani S, Igarashi Y, Tsuchikane E, Nakamura S, Seino Y, Habara M, Takeda Y, Shimoji K, Yasaka Y, Kijima M. Efficacy of drug-coated balloon angioplasty after directional coronary atherectomy for coronary bifurcation lesions (DCA/DCB registry). Catheter Cardiovasc Interv. 2021 Apr 1;97(5):E614-E623. doi: 10.1002/ccd.29185. Epub 2020 Aug 10. PMID 32776689
- [Background] Waksman R, Serra A, Loh JP, Malik FT, Torguson R, Stahnke S, von Strandmann RP, Rodriguez AE. Drug-coated balloons for de novo coronary lesions: results from the Valentines II trial. EuroIntervention. 2013 Sep;9(5):613-9. doi: 10.4244/EIJV9I5A98. PMID 24058077
- [Background] Costa MA, Kozuma K, Gaster AL, van Der Giessen WJ, Sabate M, Foley DP, Kay IP, Ligthart JM, Thayssen P, van Den Brand MJ, de Feyter PJ, Serruys PW. Three dimensional intravascular ultrasonic assessment of the local mechanism of restenosis after balloon angioplasty. Heart. 2001 Jan;85(1):73-9. doi: 10.1136/heart.85.1.73. PMID 11119468
- [Background] Yamamoto M, Hara H, Kubota S, Hiroi Y. Predictors of late lumen enlargement after drug-coated balloon angioplasty for de novo coronary lesions. EuroIntervention. 2024 May 10;20(9):602-612. doi: 10.4244/EIJ-D-23-00849. PMID 38726721
- [Background] Kleber FX, Schulz A, Waliszewski M, Hauschild T, Bohm M, Dietz U, Cremers B, Scheller B, Clever YP. Local paclitaxel induces late lumen enlargement in coronary arteries after balloon angioplasty. Clin Res Cardiol. 2015 Mar;104(3):217-25. doi: 10.1007/s00392-014-0775-2. Epub 2014 Oct 28. PMID 25349065
- [Background] Verde N, Ciliberti G, Pittorino L, Ferrone M, Franzese M, Russo M, Cioppa A, Popusoi G, Salemme L, Tesorio T, Di Gioia G. Contemporary Use of Drug-Coated Balloons for Coronary Angioplasty: A Comprehensive Review. J Clin Med. 2024 Oct 19;13(20):6243. doi: 10.3390/jcm13206243. PMID 39458193
- [Background] Jukema JW, Verschuren JJ, Ahmed TA, Quax PH. Restenosis after PCI. Part 1: pathophysiology and risk factors. Nat Rev Cardiol. 2011 Sep 13;9(1):53-62. doi: 10.1038/nrcardio.2011.132. PMID 21912414
- [Background] Whatling C, McPheat W, Hurt-Camejo E. Matrix management: assigning different roles for MMP-2 and MMP-9 in vascular remodeling. Arterioscler Thromb Vasc Biol. 2004 Jan;24(1):10-1. doi: 10.1161/01.ATV.0000100562.63144.C1. No abstract available. PMID 14707036
- [Background] Gershlick AH. Treating atherosclerosis: local drug delivery from laboratory studies to clinical trials. Atherosclerosis. 2002 Feb;160(2):259-71. doi: 10.1016/s0021-9150(01)00618-9. PMID 11849647
- [Background] Goel SA, Guo LW, Liu B, Kent KC. Mechanisms of post-intervention arterial remodelling. Cardiovasc Res. 2012 Dec 1;96(3):363-71. doi: 10.1093/cvr/cvs276. Epub 2012 Aug 22. PMID 22918976
- [Background] Fischman DL, Leon MB, Baim DS, Schatz RA, Savage MP, Penn I, Detre K, Veltri L, Ricci D, Nobuyoshi M, et al. A randomized comparison of coronary-stent placement and balloon angioplasty in the treatment of coronary artery disease. Stent Restenosis Study Investigators. N Engl J Med. 1994 Aug 25;331(8):496-501. doi: 10.1056/NEJM199408253310802. PMID 8041414
- [Background] Kastrati A, Dibra A, Mehilli J, Mayer S, Pinieck S, Pache J, Dirschinger J, Schomig A. Predictive factors of restenosis after coronary implantation of sirolimus- or paclitaxel-eluting stents. Circulation. 2006 May 16;113(19):2293-300. doi: 10.1161/CIRCULATIONAHA.105.601823. Epub 2006 May 8. PMID 16682614
- [Background] Condello F, Spaccarotella C, Sorrentino S, Indolfi C, Stefanini GG, Polimeni A. Stent Thrombosis and Restenosis with Contemporary Drug-Eluting Stents: Predictors and Current Evidence. J Clin Med. 2023 Feb 3;12(3):1238. doi: 10.3390/jcm12031238. PMID 36769886
- [Background] Madhavan MV, Kirtane AJ, Redfors B, Genereux P, Ben-Yehuda O, Palmerini T, Benedetto U, Biondi-Zoccai G, Smits PC, von Birgelen C, Mehran R, McAndrew T, Serruys PW, Leon MB, Pocock SJ, Stone GW. Stent-Related Adverse Events >1 Year After Percutaneous Coronary Intervention. J Am Coll Cardiol. 2020 Feb 18;75(6):590-604. doi: 10.1016/j.jacc.2019.11.058. PMID 32057373
- [Background] Zhong M, Tang B, Zhao Q, Cheng J, Jin Q, Fu S. Should kissing balloon inflation after main vessel stenting be routine in the one-stent approach? A systematic review and meta-analysis of randomized trials. PLoS One. 2018 Jun 27;13(6):e0197580. doi: 10.1371/journal.pone.0197580. eCollection 2018. PMID 29949587
- [Background] Gwon HC, Hahn JY, Koo BK, Song YB, Choi SH, Choi JH, Lee SH, Jeong MH, Kim HS, Seong IW, Yang JY, Rha SW, Jang Y, Yoon JH, Tahk SJ, Seung KB, Park SJ. Final kissing ballooning and long-term clinical outcomes in coronary bifurcation lesions treated with 1-stent technique: results from the COBIS registry. Heart. 2012 Feb;98(3):225-31. doi: 10.1136/heartjnl-2011-300322. Epub 2011 Sep 20. PMID 21933939
- [Background] Finet G, Derimay F, Motreff P, Guerin P, Pilet P, Ohayon J, Darremont O, Rioufol G. Comparative Analysis of Sequential Proximal Optimizing Technique Versus Kissing Balloon Inflation Technique in Provisional Bifurcation Stenting: Fractal Coronary Bifurcation Bench Test. JACC Cardiovasc Interv. 2015 Aug 24;8(10):1308-1317. doi: 10.1016/j.jcin.2015.05.016. PMID 26315733
- [Background] Ormiston JA, Webster MW, El Jack S, Ruygrok PN, Stewart JT, Scott D, Currie E, Panther MJ, Shaw B, O'Shaughnessy B. Drug-eluting stents for coronary bifurcations: bench testing of provisional side-branch strategies. Catheter Cardiovasc Interv. 2006 Jan;67(1):49-55. doi: 10.1002/ccd.20453. PMID 16003787
- [Background] Ninomiya K, Serruys PW, Garg S, Gao C, Masuda S, Lunardi M, Lassen JF, Banning AP, Colombo A, Burzotta F, Morice MC, Mack MJ, Holmes DR, Davierwala PM, Thuijs DJFM, van Klaveren D, Onuma Y; SYNTAX Extended Survival Investigators. Predicted and Observed Mortality at 10 Years in Patients With Bifurcation Lesions in the SYNTAX Trial. JACC Cardiovasc Interv. 2022 Jun 27;15(12):1231-1242. doi: 10.1016/j.jcin.2022.04.025. Epub 2022 May 17. PMID 35595676
- [Background] Lassen JF, Albiero R, Johnson TW, Burzotta F, Lefevre T, Iles TL, Pan M, Banning AP, Chatzizisis YS, Ferenc M, Dzavik V, Milasinovic D, Darremont O, Hildick-Smith D, Louvard Y, Stankovic G. Treatment of coronary bifurcation lesions, part II: implanting two stents. The 16th expert consensus document of the European Bifurcation Club. EuroIntervention. 2022 Aug 19;18(6):457-470. doi: 10.4244/EIJ-D-22-00166. PMID 35570753
- [Background] Hildick-Smith D, Arunothayaraj S, Stankovic G, Chen SL. Percutaneous coronary intervention of bifurcation lesions. EuroIntervention. 2022 Jul 22;18(4):e273-e291. doi: 10.4244/EIJ-D-21-01065. PMID 35866256
- [Background] Albiero R, Burzotta F, Lassen JF, Lefevre T, Banning AP, Chatzizisis YS, Johnson TW, Ferenc M, Pan M, Daremont O, Hildick-Smith D, Chieffo A, Louvard Y, Stankovic G. Treatment of coronary bifurcation lesions, part I: implanting the first stent in the provisional pathway. The 16th expert consensus document of the European Bifurcation Club. EuroIntervention. 2022 Aug 5;18(5):e362-e376. doi: 10.4244/EIJ-D-22-00165. PMID 35570748
- [Background] Burzotta F, Lassen JF, Louvard Y, Lefevre T, Banning AP, Daremont O, Pan M, Hildick-Smith D, Chieffo A, Chatzizisis YS, Dzavik V, Gwon HC, Hikichi Y, Murasato Y, Koo BK, Chen SL, Serruys P, Stankovic G. European Bifurcation Club white paper on stenting techniques for patients with bifurcated coronary artery lesions. Catheter Cardiovasc Interv. 2020 Nov;96(5):1067-1079. doi: 10.1002/ccd.29071. Epub 2020 Jun 24. PMID 32579300
- [Background] Lassen JF, Burzotta F, Banning AP, Lefevre T, Darremont O, Hildick-Smith D, Chieffo A, Pan M, Holm NR, Louvard Y, Stankovic G. Percutaneous coronary intervention for the left main stem and other bifurcation lesions: 12th consensus document from the European Bifurcation Club. EuroIntervention. 2018 Jan 20;13(13):1540-1553. doi: 10.4244/EIJ-D-17-00622. PMID 29061550
- [Background] Hildick-Smith D, Lassen JF, Koo BK. One or two stents for coronary bifurcation lesions? EuroIntervention. 2010 Dec;6 Suppl J:J61-4. No abstract available. PMID 21930492
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Grundeken MJ, Wykrzykowska JJ, Ishibashi Y, Garg S, de Vries T, Garcia-Garcia HM, Onuma Y, de Winter RJ, Buszman P, Linke A, Ischinger T, Klauss V, Eberli F, Corti R, Wijns W, Morice MC, di Mario C, Meier B, Juni P, Yazdani A, Copt S, Windecker S, Serruys PW. First generation versus second generation drug-eluting stents for the treatment of bifurcations: 5-year follow-up of the LEADERS all-comers randomized trial. Catheter Cardiovasc Interv. 2016 Jun;87(7):E248-60. doi: 10.1002/ccd.26344. Epub 2015 Dec 9. PMID 26649651
- [Background] Al Suwaidi J, Yeh W, Cohen HA, Detre KM, Williams DO, Holmes DR Jr. Immediate and one-year outcome in patients with coronary bifurcation lesions in the modern era (NHLBI dynamic registry). Am J Cardiol. 2001 May 15;87(10):1139-44. doi: 10.1016/s0002-9149(01)01482-5. PMID 11356386
- [Background] Steigen TK, Maeng M, Wiseth R, Erglis A, Kumsars I, Narbute I, Gunnes P, Mannsverk J, Meyerdierks O, Rotevatn S, Niemela M, Kervinen K, Jensen JS, Galloe A, Nikus K, Vikman S, Ravkilde J, James S, Aaroe J, Ylitalo A, Helqvist S, Sjogren I, Thayssen P, Virtanen K, Puhakka M, Airaksinen J, Lassen JF, Thuesen L; Nordic PCI Study Group. Randomized study on simple versus complex stenting of coronary artery bifurcation lesions: the Nordic bifurcation study. Circulation. 2006 Oct 31;114(18):1955-61. doi: 10.1161/CIRCULATIONAHA.106.664920. Epub 2006 Oct 23. PMID 17060387
- [Background] Medina A, Suarez de Lezo J, Pan M. [A new classification of coronary bifurcation lesions]. Rev Esp Cardiol. 2006 Feb;59(2):183. No abstract available. Spanish. PMID 16540043
- [Background] Lassen JF, Holm NR, Banning A, Burzotta F, Lefevre T, Chieffo A, Hildick-Smith D, Louvard Y, Stankovic G. Percutaneous coronary intervention for coronary bifurcation disease: 11th consensus document from the European Bifurcation Club. EuroIntervention. 2016 May 17;12(1):38-46. doi: 10.4244/EIJV12I1A7. PMID 27173860
- [Background] Louvard Y, Thomas M, Dzavik V, Hildick-Smith D, Galassi AR, Pan M, Burzotta F, Zelizko M, Dudek D, Ludman P, Sheiban I, Lassen JF, Darremont O, Kastrati A, Ludwig J, Iakovou I, Brunel P, Lansky A, Meerkin D, Legrand V, Medina A, Lefevre T. Classification of coronary artery bifurcation lesions and treatments: time for a consensus! Catheter Cardiovasc Interv. 2008 Feb 1;71(2):175-83. doi: 10.1002/ccd.21314. PMID 17985377
- See also: U.S. Food and Drug Administration. Medtronic Resolute Onyx Stent - Premarket Approval (PMA) — https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpma/pma.cfm?id=P160043
- See also: Sealed Envelope | Power calculator for binary outcome non-inferiority trial — https://www.sealedenvelope.com/power/binary-noninferior/